CLINICAL TRIAL: NCT00457691
Title: A Multicenter, Randomised, Double-Blind, Phase 3 Study Of Sunitinib In Metastatic Colorectal Cancer Patients Receiving Irinotecan, 5-Fluorouracil And Leucovorin (FOLFIRI) As First Line Treatment
Brief Title: Study Of FOLFIRI Chemotherapy With Or Without Sunitinib In Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6181122
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 5 fluorouracil; Drug: irinotecan; Drug: levo- leucovorin; Drug: sunitinib
- 2 (Placebo Comparator)
  Interventions: Drug: 5 fluorouracil; Drug: irinotecan; Drug: levo- leucovorin; Drug: placebo

INTERVENTIONS:
Drug: 5 fluorouracil — 400mg/m2 bolus injection day 1 followed by 2400mg/m2 continuous infusion for 46 hours every 14 days
  Arms: 1
Drug: irinotecan — 180mg/m2 iv day 1 every 14 days
  Arms: 1
Drug: levo- leucovorin — 200mg/m2 iv; day 1 every 14 days
  Arms: 1
Drug: sunitinib — 37.5mg of blinded therapy every day for 28 days followed by 14 days of blinded therapy free period
  Arms: 1
Drug: 5 fluorouracil — 400mg/m2 bolus injection day 1 followed by 2400mg/m2 continuous infusion for 46 hours every 14 days
  Arms: 2
Drug: irinotecan — 180mg/m2 iv day 1 every 14 days
  Arms: 2
Drug: levo- leucovorin — 200mg/m2 iv; day 1 every 14 days
  Arms: 2
Drug: placebo — 37.5mg of blinded placebo therapy every day for 28 days followed by 14 days of blinded therapy free period
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of FOLFIRI (Irinotecan, Leucovorin and 5 Fluorouracil) chemotherapy when combined with sunitinib or FOLFIRI chemotherapy without adding sunitinib as the first line treatment of patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
On June 25, 2009, the independent Data Monitoring Committee (DMC) reviewed the progress of Study A6181122. The DMC determined Study A6181122 had met pre-specified futility criteria and was unlikely to meet its primary endpoint to demonstrate a statistically significant improvement in progression-free survival (PFS) in patients treated with sunitinib plus FOLFIRI versus placebo plus FOLFIRI. No new safety findings were noted. Pfizer notified clinical trial investigators involved in the study and regulatory agencies of these findings. Patients receiving benefit on treatment as determined by the investigator may remain on study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed (histologically or cytologically) colorectal adenocarcinoma with metastatic disease.
* Not received previous therapy for metastatic colorectal disease but for whom FOLFIRI treatment is clinically indicated.
* Adequate organ function defined by blood test.

Exclusion Criteria:

* History of another primary cancer in the last 3 years.
* Previous full field radiotherapy within the last 4 weeks or limited field radiotherapy within 2 weeks of enrolling into the study. Or previous radiation treatment of more that 30% of the bone marrow.
* History of presence of brain metastasis, spinal cord compression carcinomatous meningitis or leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (109):
- Argentina (2):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Santa Fe, Santa Fe Province
- Australia (4):
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, East Bentleigh, Victoria
  - Pfizer Investigational Site, Frankston, Victoria
  - Pfizer Investigational Site, Fremantle, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Sankt Pölten
  - Pfizer Investigational Site, Vienna
- Belgium (4):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- Brazil (4):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Santo André, São Paulo
- Bulgaria (5):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Rousse
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
  - Pfizer Investigational Site, Varna
- Canada (2):
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
- Pfizer Investigational Site, Santiago, RM, Chile
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Pasto, Departamento de Nariño
- Pfizer Investigational Site, Nicosia, Cyprus
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Příbram
- Germany (9):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Esslingen am Neckar
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Mönchengladbach
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Regensburg
- Hong Kong (3):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Tuen Mun, New Territories
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
- India (4):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Vellore, Tamil Nadu
- Ireland (2):
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Mexico (3):
  - Pfizer Investigational Site, Acapulco de Juárez, Guerrero
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Ciudad Obregón, Sonora
- Norway (2):
  - Pfizer Investigational Site, Førde
  - Pfizer Investigational Site, Tønsberg
- Pfizer Investigational Site, Warsaw, Poland
- Portugal (3):
  - Pfizer Investigational Site, Evora
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Santa Maria da Feira
- Pfizer Investigational Site, Cluj-Napoca, Cluj, Romania
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Serbia (4):
  - Pfizer Investigational Site, Belgrade, Serbia
  - Pfizer Investigational Site, Kamenitz, Serbia
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Kamenitz
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Pfizer Investigational Site, Bratislava, Slovakia
- South Africa (5):
  - Pfizer Investigational Site, Observatory
  - Pfizer Investigational Site, Panorama
  - Pfizer Investigational Site, Parktown
  - Pfizer Investigational Site, Port Elizabeth
  - Pfizer Investigational Site, Sandton
- South Korea (4):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
- Spain (8):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Móstoles, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Zaragoza, Zaragoza
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- Taiwan (8):
  - Pfizer Investigational Site, Kaohsiang Hsien, Taiwan
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Chiayi County
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Kwei-Shan, Taoyuan
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Thailand (4):
  - Pfizer Investigational Site, Rachathevee, Bangkok
  - Pfizer Investigational Site, Muang, Changwat Khon Kaen
  - Pfizer Investigational Site, Muang, Chiang Mai
  - Pfizer Investigational Site, Bangkok
- Ukraine (5):
  - Pfizer Investigational Site, Cherkasy
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Uzhhorod
- United Kingdom (3):
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Carrato A, Swieboda-Sadlej A, Staszewska-Skurczynska M, Lim R, Roman L, Shparyk Y, Bondarenko I, Jonker DJ, Sun Y, De la Cruz JA, Williams JA, Korytowsky B, Christensen JG, Lin X, Tursi JM, Lechuga MJ, Van Cutsem E. Fluorouracil, leucovorin, and irinotecan plus either sunitinib or placebo in metastatic colorectal cancer: a randomized, phase III trial. J Clin Oncol. 2013 Apr 1;31(10):1341-7. doi: 10.1200/JCO.2012.45.1930. Epub 2013 Jan 28. PMID 23358972
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181122&StudyName=Study%20Of%20FOLFIRI%20Chemotherapy%20With%20Or%20Without%20Sunitinib%20In%20Patients%20With%20Metastatic%20Colorectal%20Cancer%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRI + Sunitinib: Intravenous (IV) irinotecan (180 milligrams per square meter [mg/m²]), and levo-leucovorin (200 mg/m² or leucovorin at 400 mg/m²) immediately followed by 5-fluorouracil (5-FU) IV bolus (400 mg/m²) and 5-FU 46-hour continuous IV infusion (2400 mg/m²) every 2 weeks (FOLFIRI). Sunitinib 37.5 mg oral capsules once daily on Schedule 4/2 (4 weeks on, 2 weeks off). Three courses of FOLFIRI were administered during every 6 week sunitinib cycle.
- FOLFIRI + Placebo: IV irinotecan (180 mg/m²), and levo-leucovorin (200 mg/m² or leucovorin at 400 mg/m²) immediately followed by 5-FU IV bolus (400 mg/m²) and 5-FU 46-hour continuous IV infusion (2400 mg/m²) every 2 weeks (FOLFIRI). Placebo oral capsules once daily on Schedule 4/2 (4 weeks on, 2 weeks off). Three courses of FOLFIRI were administered during every 6 week placebo cycle.
Period: Overall Study
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Started | 386 | 382
Completed | 0 | 0
Not Completed | 386 | 382
Not completed — Adverse Event | 4 | 1
Not completed — Death | 163 | 148
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 23 | 14
Not completed — Study terminated by Sponsor | 1 | 1
Not completed — Subject refused (reason other than AE) | 14 | 19
Not completed — Disease progression, study terminated | 180 | 196

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo | Total
Number analyzed (Participants) | 386 | 382 | 768
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.36) | 57.6 (10.77) | 58.1 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 179 | 343
  Male | 222 | 203 | 425

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS defined as time from date of randomization to date of first documentation of objective tumour progression or death due to any cause, whichever occurred first.
Time Frame: First dose of study treatment up to 30 months
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Weeks | 33.6 [30.80 to 36.60] | 36.6 [32.90 to 40.00]
Statistical Analysis 1: Comparison: FOLFIRI + Sunitinib vs FOLFIRI + Placebo; Test type: Superiority or Other; p = 0.8072, Log Rank — p-value from 1-sided log-rank test, stratified by Eastern Cooperative Oncology Group (ECOG) performance status, organ sites with disease, primary tumor site, prior adjuvant treatment; Hazard Ratio (HR) = 1.095, 95% CI 2-sided [0.892 to 1.344]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. OS data were censored on the day following the date of the last contact at which the patient was known to be alive.
Time Frame: Baseline up to 30 months
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Weeks | 87.9 [75.20 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored events | 85.9 [81.10 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored events
Statistical Analysis 1: Comparison: FOLFIRI + Sunitinib vs FOLFIRI + Placebo; Test type: Superiority or Other; p = 0.9163, Log Rank — p-value from 1-sided log-rank test, stratified by ECOG performance status, organ sites with disease, primary tumor site, prior adjuvant treatment; Hazard Ratio (HR) = 1.171, 95% CI 2-sided [0.936 to 1.466]

3. Secondary Outcome: Number of Participants With Overall Confirmed Objective Response
Description: Objective disease response: participants with a confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions. PR was defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1 up to 30 months
Measure: Number; unit: Participants
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Participants | 124 | 128

4. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first objective documentation of CR or PR that was subsequently confirmed to the first documentation of disease progression or to death due to any cause, whichever occurred first.
Time Frame: Day 28 of Cycle 1 up to 30 months
Population: ITT Population (participants with a confirmed objective tumor response).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 124 | 128
Weeks | 30.1 [27.10 to 37.20] | 39.0 [31.90 to 49.00]

5. Secondary Outcome: Change From Baseline in Monroe Dunaway (MD) Anderson Symptom Assessment Inventory of Gastrointestinal Symptoms (MDASI-GI) Symptom Intensity Score
Description: Symptom Intensity score is comprised of the sum of 13 MDASI core items (ie, pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, remembering things, lack of appetite, drowsiness, dry mouth, sadness, vomiting, numbness or tingling). Participant asked to rate severity of each symptom at their worst in past 24 hours; each item rated from 0 to 10, with 0=symptom not present and 10=as bad as you can imagine; lower scores indicated better outcome (range: 0 to 130).
Time Frame: Day 1 of Cycles 1-3 and Day 1 of every odd-numbered cycle thereafter until end of treatment (EOT)/withdrawal
Population: ITT population. The change from baseline MDASI-GI within each treatment arm was evaluated only for those cycles where at least 10 participants had available data (Cycles 2, 3, 5, 7, 9, and 11).
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Scores on a scale
  Cycle 2, Day 1 | 1.7 [-0.4 to 3.8] | 0.4 [-1.3 to 2.2]
  Cycle 3, Day 1 | 0.8 [-1.4 to 2.9] | 0.9 [-1.1 to 3.0]
  Cycle 5, Day 1 | 1.0 [-1.6 to 3.7] | 1.8 [-0.4 to 3.9]
  Cycle 7, Day 1 | 0.7 [-2.6 to 4.0] | 2.7 [-0.3 to 5.7]
  Cycle 9, Day 1 | 0.8 [-5.6 to 7.1] | 1.2 [-3.3 to 5.6]
  Cycle 11, Day 1 | 5.0 [-3.2 to 13.2] | -2.7 [-8.4 to 3.0]

6. Secondary Outcome: Change From Baseline in MDASI-GI Symptom Interference Score
Description: Symptom Interference score is comprised of the sum 6 function items from MDASI core (general activity, walking, work, mood, relations with other people, and enjoyment of life). Participant asked to rate how much symptoms have interfered in past 24 hours; each item rated from 0 to 10, with 0=did not interfere and 10=interfered completely; lower scores indicated better outcome (range: 0 to 60).
Time Frame: Day 1 of Cycles 1-3 and Day 1 of every odd-numbered cycle thereafter until EOT/withdrawal
Population: ITT population. The change from baseline MDASI-GI within each treatment arm was evaluated only for those cycles where at least 10 participants had available data (Cycles 2, 3, 5, 7, 9, 11).
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
scores on a scale
  Cycle 2, Day 1 | 0.0 [-1.4 to 1.4] | -1.3 [-2.6 to 0.0]
  Cycle 3, Day 1 | -0.1 [-1.8 to 1.6] | -1.7 [-3.2 to -0.2]
  Cycle 5, Day 1 | 0.2 [-1.8 to 2.1] | -1.2 [-3.1 to 0.6]
  Cycle 7, Day 1 | -0.5 [-2.9 to 1.9] | -0.2 [-2.7 to 2.3]
  Cycle 9, Day 1 | 2.1 [-0.7 to 4.9] | -1.7 [-4.7 to 1.2]
  Cycle 11, Day 1 | 3.1 [-1.2 to 7.4] | -1.0 [-6.5 to 4.5]

7. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) EQ-5D Self-Report Questionnaire
Description: EQ-5D: participant-rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problem); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain. Score is transformed and results in total score range -1.11 to 1.000; higher score indicates better health state.
Time Frame: Day 1 of Cycles 1-3 and Day 1 of every odd-numbered cycle thereafter until EOT/withdrawal
Population: ITT population. The EQ-5D health state index results were assessed for only those cycles where at least 10 participants on either treatment arm had available data (Cycles 2, 3, 5, 7, 9, and 11).
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Scores on a scale
  Cycle 2, Day 1 | 0.02 [0.00 to 0.04] | 0.04 [0.02 to 0.05]
  Cycle 3, Day 1 | 0.02 [0.00 to 0.04] | 0.04 [0.02 to 0.06]
  Cycle 5, Day 1 | 0.02 [-0.00 to 0.05] | 0.03 [0.01 to 0.05]
  Cycle 7, Day 1 | 0.03 [-0.01 to 0.06] | 0.05 [0.02 to 0.07]
  Cycle 9, Day 1 | 0.00 [-0.05 to 0.05] | 0.05 [0.02 to 0.08]
  Cycle 11, Day 1 | 0.01 [-0.04 to 0.06] | 0.09 [0.05 to 0.14]

8. Secondary Outcome: Change From Baseline in EuroQol (EQ) Visual Analog Scale (VAS) (EQ-VAS)
Description: EQ-5D: participant-rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Day 1 of Cycles 1-3 and Day 1 of every odd-numbered cycle thereafter until EOT/withdrawal
Population: ITT population. The change from baseline scores for EQ-VAS were assessed for only those cycles where at least 10 participants on either treatment arm had available data (Cycles 2, 3, 5, 7, 9, and 11).
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Number analyzed (Participants) | 386 | 382
Scores on a scale
  Cycle 2, Day 1 | 1.0 [-1.1 to 3.0] | 3.3 [1.3 to 5.3]
  Cycle 3, Day 1 | 1.7 [-0.7 to 4.0] | 4.3 [2.0 to 6.6]
  Cycle 5, Day 1 | 1.8 [-0.6 to 4.1] | 6.6 [3.5 to 9.8]
  Cycle 7, Day 1 | 3.8 [-0.4 to 8.1] | 4.3 [0.4 to 8.2]
  Cycle 9, Day 1 | -0.9 [-6.2 to 4.5] | 4.0 [-0.5 to 8.5]
  Cycle 11, Day 1 | -1.6 [-6.7 to 3.6] | 9.0 [2.6 to 15.3]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | FOLFIRI + Sunitinib | FOLFIRI + Placebo
Serious Adverse Events (participants affected / at risk) | 170/384 | 111/379
Other Adverse Events (participants affected / at risk) | 382/384 | 362/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI + Sunitinib (N=384) | FOLFIRI + Placebo (N=379)
Anaemia (Blood and lymphatic system disorders) | 9 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 11
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 3
Neutropenia (Blood and lymphatic system disorders) | 26 | 6
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Pupils unequal (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Colonic obstruction (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 23 | 19
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrooesophagitis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 8
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 8 | 10
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 11
Asthenia (General disorders) | 3 | 4
Catheter related complication (General disorders) | 0 | 1
Catheter thrombosis (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 1
Death (General disorders) | 4 | 4
Disease progression (General disorders) | 12 | 3
Fatigue (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 17 | 12
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 3 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 4 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Implant site cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Liver abscess (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 7
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pseudomonas pseudomallei infection (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Renal function test abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukoerythroblastosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 3 | 3
Hydroureter (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Immobile (Social circumstances) | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 3
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI + Sunitinib (N=384) | FOLFIRI + Placebo (N=379)
Anaemia (Blood and lymphatic system disorders) | 120 | 74
Leukopenia (Blood and lymphatic system disorders) | 107 | 49
Neutropenia (Blood and lymphatic system disorders) | 315 | 188
Thrombocytopenia (Blood and lymphatic system disorders) | 129 | 21
Abdominal distension (Gastrointestinal disorders) | 21 | 26
Abdominal pain (Gastrointestinal disorders) | 89 | 73
Abdominal pain upper (Gastrointestinal disorders) | 43 | 28
Constipation (Gastrointestinal disorders) | 89 | 72
Diarrhoea (Gastrointestinal disorders) | 247 | 182
Dyspepsia (Gastrointestinal disorders) | 45 | 24
Nausea (Gastrointestinal disorders) | 190 | 181
Stomatitis (Gastrointestinal disorders) | 88 | 45
Vomiting (Gastrointestinal disorders) | 144 | 129
Asthenia (General disorders) | 70 | 65
Chest pain (General disorders) | 28 | 9
Fatigue (General disorders) | 120 | 93
Mucosal inflammation (General disorders) | 87 | 66
Oedema peripheral (General disorders) | 27 | 26
Pyrexia (General disorders) | 67 | 53
Upper respiratory tract infection (Infections and infestations) | 24 | 20
Alanine aminotransferase increased (Investigations) | 23 | 12
Aspartate aminotransferase increased (Investigations) | 22 | 9
Weight decreased (Investigations) | 36 | 17
Decreased appetite (Metabolism and nutrition disorders) | 116 | 82
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 32
Dizziness (Nervous system disorders) | 29 | 27
Dysgeusia (Nervous system disorders) | 30 | 20
Headache (Nervous system disorders) | 44 | 28
Insomnia (Psychiatric disorders) | 55 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 | 21
Alopecia (Skin and subcutaneous tissue disorders) | 128 | 121
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 77 | 26
Rash (Skin and subcutaneous tissue disorders) | 41 | 32
Skin discolouration (Skin and subcutaneous tissue disorders) | 22 | 2
Hypertension (Vascular disorders) | 56 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.